CLINICAL TRIAL: NCT05842850
Title: Increased Risk of Non-alcoholic Fatty Liver Disease in Low Birth Weight Individuals - Reversibility and Mechanistic Studies.
Brief Title: Non-alcoholic Fatty Liver Disease in Low Birth Weight Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Aarhus University Hospital (Other); Lund University (Other)
Responsible Party: Principal Investigator, Charlotte Brøns, Principal investigator, Steno Diabetes Center Copenhagen
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NAFLD reversibility
Record Dates: First submitted 2023-04-11; First posted 2023-05-06 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: NAFLD
Keywords: Adipose tissue biology; Caloric restriction; Insulin resistance; Energy expenditure; Insulin secretion
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Participants will be recruited from a nested case-control (NAFLD) screening study. Participants will be examined on two separate days at baseline (both groups) and after 4-weeks caloric restriction (LBW with NAFLD only). The caloric restriction intervention will start immediately after completion of baseline examinations. Participants will adhere to a caloric restriction protocol for 4-weeks limiting daily food intake to a window of 8 hours (8am to 4pm) and water-fasting for the remaining hours of the day. Participants will be instructed to eat a balanced diet according to the current dietary guidelines reduced by 20% calories to ensure energy deficit. A weighed food diary and accelerometers will be used for 3-days to estimate baseline dietary intake and physical activity and to monitor intervention adherence after 2 and 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LBW individuals with NAFLD (Experimental): LBW individuals with NAFLD
  Interventions: Behavioral: Caloric restriction intervention
- NBW controls without NAFLD (Placebo Comparator): Age-, gender- and body mass index-matched NBW controls without NAFLD
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Caloric restriction intervention — The intervention consist of 4-weeks limiting daily food intake to a window of 8 hours (8am to 4pm) and water-fasting for the remaining hours of the day. Participants (LBW NAFLD individuals only) will be instructed to eat a balanced diet according to the current dietary guidelines reduced by 20% calories to ensure energy deficit.
  Other Names: No intervention
  Arms: LBW individuals with NAFLD
Other: No intervention — No intervention
  Arms: NBW controls without NAFLD

SUMMARY:
The investigators will conduct a proof-of-principle deep phenotyping 4-weeks caloric restriction intervention study in low birth weight (LBW) subjects with NAFLD and normal birth weight (NBW) controls. Furthermore, the investigators will provide extended in-depth mechanistic insight into the role of impaired subcutaneous adipose tissue (SAT) expandability in ectopic fat deposition in LBW subjects in LBW individuals with and without NAFLD.

DETAILED DESCRIPTION:
An adverse fetal environment characterized by low birth weight (LBW) plays a key role in the development of type 2 diabetes (T2D). The investigators recently demonstrated a 3-fold increase in liver fat in 26 early middle-aged LBW compared to 22 normal birth weight (NBW) men, and 20% of the LBW - but none of the normal birth weight (NBW) - men had previously unknown non-alcoholic fatty liver disease (NAFLD). The investigators hypothesize that ectopic fat deposition and NAFLD is among the earliest disease manifestations and on the critical path to the development of more severe cardiometabolic disease in LBW. The investigators furthermore hypothesize, that LBW individuals exhibit ectopic liver fat due to reduced capacity to store fat in the subcutaneous adipose tissue (SAT) depot, and that early detection and subsequent intensive caloric restriction, in middle-aged LBW individuals with overt NAFLD, may represent a targeted and highly efficient way forward to prevent more severe cardiometabolic disease manifestations in LBW subjects. To further explore the recent findings, the investigators aim to perform an extended nested case-control screening study for NAFLD in 250 early middle-aged non-obese LBW men and women, and subsequently to conduct a deep-phenotyping, proof-of-principle 4 week time-restricted eating (TRE) intervention study in 12 LBW subjects with NAFLD including measures of hepatic fat content, glucose, insulin and lipid metabolism, as well as 24h metabolic profiles using respiratory chambers. Finally, the investigators will provide extended in-depth mechanistic insight into transcriptional, epigenetic as well as functional SAT and preadipocyte perturbations underlying impaired SAT expandability in LBW individuals with and without NAFLD and NBW controls studied before and after different dietary interventions including TRE and high carbohydrate overfeeding.

ELIGIBILITY:
Inclusion Criteria:

* LBW subjects with NAFLD (liver fat content ≥5% liver fat content verified on MRS)
* Gender- and body mass index-matched NBW controls without NAFLD
* Born at term (weeks 39-41)

Exclusion Criteria:

* BMI<18.5 and BMI>30 kg/m2
* Family history of diabetes (siblings, parent, and grandparents)
* Disease/medication known to affect primary outcome
* Self-reported high physical activity level
* Alcohol intake above general recommendations.
* Metabolic/liver disease
* Weight gain/loss of >3 kg within the past 6 months

Ages: 35 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Liver fat content | Change from baseline in liver fat content at 4 weeks
  Liver elastography (FibroScan)
Liver fat content | Change from baseline in liver fat content at 4 weeks
  Validation by Magnetic resonance spectroscopy (MRS)

SECONDARY OUTCOMES:
Liver fibrosis | Baseline and after 4 weeks
  Liver elastography (FibroScan)
Whole-body insulin sensitivity | Baseline and after 4 weeks
  Stepwise hyperinsulinemic-euglycemic clamp
Beta-cell function | Baseline and after 4 weeks
  Intravenous glucose tolerance test
Glucose turnover rate | Baseline and after 4 weeks
  Stable isotope dilution technique
Fat turnover rate | Baseline and after 4 weeks
  Stable isotope dilution techniques
Urea turnover rate | Baseline and after 4 weeks
  Stable isotope dilution techniques
24-hour energy metabolism | Baseline and after 4 weeks
  Indirect calorimetry in respiratory chamber
Body composition | Baseline and after 4 weeks
  DEXA scan

OTHER OUTCOMES:
Adipocyte size | Baseline and after 4 weeks
  Adipose tissue immunohistochemistry
Collagen content | Baseline and after 4 weeks
  Adipose tissue immunohistochemistry
Transcriptomics | Baseline and after 4 weeks
  RNAseq of bulk subcutaneous adipose tissue
Transcriptomics | Baseline and after 4 weeks
  RNAseq of ex vivo cultured preadipocytes
Epigenetics | Baseline and after 4 weeks
  Genome-wide DNA methylation of subcutaneous adipose tissue
Epigenetics | Baseline and after 4 weeks
  Genome-wide DNA methylation of ex vivo cultured preadipocytes
Metabolism of ex vivo differentiated preadipocytes | Baseline and after 4 weeks
  Functional characterization of lipid metabolism
Metabolism of ex vivo differentiated preadipocytes | Baseline and after 4 weeks
  Functional characterization of glucose metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Brøns, PhD, Principal Investigator — Steno Diabetes Center Copenhagen

IPD SHARING:
Plan to Share IPD: No